CLINICAL TRIAL: NCT05212740
Title: Oral Corticosteroids Versus Exercises On Treatment Of Frozen Shoulder,
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Zeynal YASACI, Research Assistant; Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Istanbul Unıversity-Cerrahpasa
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Frozen Shoulder
Keywords: frozen shoulder; adhesive capsulitis; corticosteroid; exercise
MeSH Terms: conditions — Bursitis; Motor Activity | interventions — Adrenal Cortex Hormones; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid (Experimental): The participants will receive prednisolone for four weeks.
  Interventions: Drug: Corticosteroid
- Exercise (Active Comparator): The participants will receive joint mobilization techniques, stretching and home exercise.
  Interventions: Other: Exercise

INTERVENTIONS:
Drug: Corticosteroid — The treatment will initiate with a dose of 0.5 mg/kg/day prednisolone for two weeks and the dose will halve in the next two weeks.
  Arms: Corticosteroid
Other: Exercise — The exercise program will be performed two times per week for six weeks for 12 sessions.
  Arms: Exercise

SUMMARY:
The purpose of this study is to compare the efficacy of exercise and oral corticosteroids the treatment of a FS.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed and meet the inclusion criteria will be randomized a double blind manner in a 1:1 (participant and investigator) to oral corticosteroids or exercise.

ELIGIBILITY:
Inclusion Criteria:

1. between ages 18-60 years
2. loss of passive motion of the glenohumeral joint greater than 25% or 30 in at least 2 directions (flexion, external rotation, and internal rotation) compared with the contralateral side
3. The pain VAS more than 7 (10 in total)

Exclusion Criteria:

1. bilateral frozen shoulder
2. rotator cuff tear
3. previous corticosteroid injection at the affected shoulder within 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in function on DASH at 6th and 12th week | Baseline,6th week and 12th week
  The DASH is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.

SECONDARY OUTCOMES:
Change from baseline in function on ASES at 6th and 12th week | Baseline,6th week and 12th week
  The ASES score is a 10-item measure of shoulder pain and function. Pain is assessed on a 10-cm visual analog scale (VAS) and accounts for 50% of the total score. The remaining 50% of the score is determined by the responses to 10 4-point Likert-scale questions related to physical function.
Change from baseline in range of motion (ROM) at 6th and 12th week | Baseline,6th week and 12th week
  The joint's range of motion is the distance that the joint can extend.
Change from baseline in depression and anxiety on HADS at 6th and 12th week | Baseline,6th week and 12th week
  HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression. HADS scoring was done before and after low-vision consultation to see whether there was a change in the scoring.
Change from baseline in pain on VAS at 6th and 12th week | Baseline,6th week and 12th week
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Çelik, Study Director — Istanbul University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Faculty Medicine, Istanbul, Fatih
  - İÜC Sağlık Bilimleri Fakültesi, Istanbul